CLINICAL TRIAL: NCT06922058
Title: The Use of Virtual Reality Glasses to Reduce Anxiety in Fixed Orthodontic Treatments
Brief Title: The Use of Virtual Reality Glasses to Reduce Anxiety in Fixed Orthodontic Treatments in Children Aged 10-15 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Fatma Betül Yucel, Principal Investigator, Biruni University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-KAEK-79-23-11
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Anxiety
Keywords: Virtual reality; orthodontics; anxiety; pulse oximeter; visual analog scale; STAI; CASI
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients treated with VR glasses (Experimental): These patients are asked anxiety tests before and after the treatment. They are watching animation on VR glasses during the first day of the treatment. Their values are recording by pulse-oximetry.
  Interventions: Device: Virtual Reality Glasses
- Patients treated without VR glasses (No Intervention): These patients are asked anxiety tests before and after treatment. Their values are recording by pulse-oximetry.

INTERVENTIONS:
Device: Virtual Reality Glasses — Virtual reality glasses haven't used in orthodontics in another clinical study.
  Arms: Patients treated with VR glasses

SUMMARY:
This study aims to manage anxiety and fear experienced by young patients during orthodontic treatments through the use of virtual reality glasses, ensuring a more comfortable procedural experience.

The study included twenty-six patients who visited the faculty of dentistry. Thirteen patients in the study group were shown animation through virtual reality glasses during the procedure. The 13 patients in the control group underwent standard treatment procedures without virtual reality glasses. Both groups were asked questions from the CASI and Trait Anxiety Inventory at the beginning of the procedure, State Anxiety Inventory at the beginning and at the end of the procedure, and pulse rate, saturation and VAS values were recorded.

The implementation of virtual reality glasses in orthodontic treatments has been shown to effectively manage anxiety by distracting patients from what is actually happening.

This study shows that virtual reality goggles reduce the anxiety experienced by patients during orthodontic treatment. These results offer a different treatment process that can increase treatment comfort in clinical practice.

DETAILED DESCRIPTION:
Orthodontic treatments are treatments that have less knowledge and experience among patients compared to other dental procedures, and therefore have a more uncertain process for patients. The tools and materials used in orthodontic treatments also differ from the materials that patients are familiar with using in other dental procedures. Patients aged 10-15 years were identified as an age group in which fixed orthodontic treatment could be started for the age range of our study group, who had less experience in dental treatments compared to adults, and therefore the level of anxiety was mostly higher. In addition, it has been observed that the bracket placement session, which is the first session of fixed orthodontic treatment, is longer than the sessions in which other orthodontic procedures are performed, and during this period, patients in the age group we have chosen tend to question the remaining time and want to check their mobile phones, and it is believed that virtual reality (VR) glasses can be utilized to enhance the comfort of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children who needed and accepted fixed orthodontic treatment,
* Children who had not received orthodontic treatment before
* Children who did not have any psychiatric or systemic disorders

Exclusion Criteria:

* Children who had previously undergone orthodontic treatment
* Children with psychiatric or systemic disorders.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Pulse | 1 hour
  Throughout the session, pulse levels were recorded using a pulse oximeter at three points: before, during, and after the session.
  The normal pulse rate is between 60-100 beats/minute in children and adolescents aged 11-17 years. In our study, the values obtained in measurements made according to time were compared with each other.
Oxygen Saturation | 1 hour
  Throughout the session, saturation levels were recorded using a pulse oximeter at three points: before, during, and after the session.
  Oxygen saturation in children is within the normal range when read between 94-100%. In our study, the data obtained in measurements made according to time were compared with each other.

SECONDARY OUTCOMES:
Visual Analog Scale | 1 hour
  Patients rated their anxiety levels on the Visual Analog Scale (VAS) before and at the end of the session. On the scale, it can be scored between 1 and 10. 1 represents the lowest level of anxiety and 10 represents the highest level of anxiety.
Stait-Trait Anxiety Scale | 1 hour
  Before and after the session, patients were asked the questions of stait-trait anxiety scale.
  In the State Anxiety Scale, the answer options are (1) Never, (2) A little, (3) A lot and (4) Completely; the options in the Trait Anxiety Scale are (1) Almost never, (2) Sometimes, (3) Very often and (4) Almost always.
  There are two types of statements in the scales: Direct expressions express negative emotions; reversed expressions express positive emotions. When scoring these second type of statements, those with a weight value of 1 turn into 4 and those with a weight value of 4 turn into 1. In direct statements, answers with a value of 4 indicate that anxiety is high. In reversed statements, answers with a value of 1 indicate high anxiety. The scores obtained from both scales theoretically range between 20 and 80.High scores indicate a high level of anxiety and low scores indicate a low level of anxiety.The average score level determined in the applications varies between 36 and 41.
Children Anxiety Sensitivity Index | 1 hour
  Patients were assessed using the Children Anxiety Sensitivity Index before the session.
  It is an eighteen-item self-report scale. It questions children's feelings after internal and external stimuli that may cause anxiety.
  It is organised as a 3-point Likert-type scale. It is scored as not at all (1), a little (2), very much (3), which can be easily understood even by children as young as 7 years old. The minimum score is 18, the maximum score is 54. Low scores indicate low anxiety, high scores indicate high anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Aslı Konca Taşova, Assistant Professor, Study Director — Uskudar University
Locations (1):
- Biruni University Dentistry Faculty Departments of Orthodontics, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared on reasonable request to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending a year after the publication of results.
Access Criteria: The investigators can access to the corresponding author by e-mail.